CLINICAL TRIAL: NCT04086446
Title: A Randomized Clinical Trial of Transcranial Direct Current Stimulation(tDCS) Treatment for Drug-naïve Obsessive-Compulsive Disorder(OCD)
Brief Title: Transcranial Direct Current Stimulation (tDCS) in the Treatment of Drug-naïve Obsessive-compulsive Disorder(OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-004
Record Dates: First submitted 2019-09-08; First posted 2019-09-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS (Active Comparator): Cathode transcranial direct current stimulation over the right OFC will be applied once a day, 5 days a week, for 2 weeks.
  Interventions: Device: high-definition transcranial direct current stimulation
- sham tDCS (Sham Comparator): The sham transcranial direct current stimulation over the right OFC will be applied once a day, 5 days a week, for 2 weeks.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: high-definition transcranial direct current stimulation — The tDCS device will deliver a direct current of 1.5mA during 20 minutes. Cathode electrode will be localized in front of the right OFC on the Fp2 point according to the EEG international reference. Four anode electrodes will be placed around FP2 (i.e. Fpz, AFz, AF4, AF8)
  Arms: active tDCS
Device: Sham tDCS — The same procedure will be applied except that the tDCS device will only deliver a current stimulation for the first and last 15 seconds.
  Arms: sham tDCS

SUMMARY:
This study will evaluate the possible therapeutic effects of Transcranial Direct Current Stimulation (tDCS) in drug-naïve obsessive-compulsive disorder (OCD) patients, and the underlying neural mechanism by magnetic resonance imaging (MRI),transcranial magnetic stimulation and electroencephalography (TMS-EEG).

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy of tDCS over orbitofrontal cortex (OFC) in treatment of drug-naïve OCD patients. 60 drug-naïve OCD patients will be randomized into two groups (i.e. active or sham stimulation). tDCS stimulation will be performed once a day, five times a week, for two weeks. The investigators will assess symptom severity before and after two weeks of tDCS. Through the study, Yale-Brown Obsessive Compulsive Scale（Y-BOCS）, the Obsessive Compulsive Inventory-Revised (OCI-R), the Beck Depression Inventory (BDI), the Beck Anxiety Inventory (BAI), Perceived Stress Scale (PSS), Pittsburgh sleep quality index (PSQI)and side-effect questionnaire will be obtained by a trained investigator. The patients will also receive MRI scan and TMS-EEG.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-50 years old;
* DSM-5 criteria for OCD;
* Y-BOCS total score > or = 16, discontinued medication for at least 8 weeks before tDCS stimulation.
* >or＝9 years education

Exclusion Criteria:

* Any axis I psychiatric disorder comorbidity
* The inability to receive tDCS because of metallic implants, or history of seizures，or 3.history of head injury, or history of neurosurgery.
* Participants with claustrophobic, heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.
* Any current significant medical condition.
* serious suicide risk

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale(Y-BOCS) score | Up to 3 months
  It assesses the severity of OCD symptoms. The Y-BOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.The responder on Y-BOCS is defined as a Y-BOCS decrease at least 35% from the baseline at post-treatment.

SECONDARY OUTCOMES:
Change in Obsessive Compulsive Inventory-Revised(OCI-R) | Up to 3 months
  It is an inventory of OCD symptoms with 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Change in Beck Depression Inventory(BDI) | Up to 3 months
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in Beck Anxiety Inventory (BAI) | Up to 3 months
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Change in Perceived Stress Scale(PSS) | Up to 3 months
  It is a 10-item, 5-point Likert scale(0 to 4) to measure the degree to which situations in one's life are appraised as stressful.The total score ranges from 0 to 40, with lower total scores representing a better outcome.
Change in Pittsburgh sleep quality index(PSQI) | Up to 3 months
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Change in Side-effect questionnaire | Up to 3 months
  It consists of 10-item and uses 0 to 3 severity scale to rate the intensity of side effects. Total scores range from 0 to 30, with higher scores indicating more severe side-effect. It also assesses the relation between side-effect and the effects of tDCS using 0 to 4 scale. Total scores range from 0 to 40, with higher score indicating the greater relation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No